CLINICAL TRIAL: NCT01231568
Title: An Open-Label Study to Examine the Effects of a High-Fat Meal and Particle Size on the Pharmacokinetics of Orally Administered GSK2118436 in Subjects With BRAF Mutation-Positive Tumor
Brief Title: An Open Label Study to Examine the Effects of a High-Fat Meal and Particle Size on the Pharmacokinetics of Orally Administered GSK2118436 in Subjects With BRAF Mutation Positive Tumor
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 113468
Record Dates: First submitted 2010-10-21; First posted 2010-11-01 (Estimated); Last update posted 2017-11-14 (Actual); Status verified 2017-11

CONDITIONS: Cancer
Keywords: food effect; high fat meal; GSK2118436; pharmacokinetic; particle size; BRAF inhibitor; BRAF positive tumor
MeSH Terms: conditions — Neoplasms | interventions — OOS-A regimen; Regimen B

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Cohort 1 Treatment Sequence 1 (Experimental): Subjects will receive two 75 mg micronized gelatin capsules, dosed fasted (Regimen A) in Period 1 and two 75 mg non-micronized gelatin capsules, dosed fasted (Regimen B) in Period 2. Dosing will occur in the morning of Day 1 in each period, and dosing between periods will be separated by at least one week.
  Interventions: Drug: Regimen A; Drug: Regimen B
- Cohort 1 Treatment Sequence 2 (Experimental): Subjects will receive two 75 mg non-micronized gelatin capsules, dosed fasted (Regimen B) in Period 1 and two 75 mg micronized gelatin capsules, dosed fasted (Regimen A) in Period 2. Dosing will occur in the morning of Day 1 in each period, and dosing between periods will be separated by at least one week.
  Interventions: Drug: Regimen A; Drug: Regimen B
- Cohort 2 Treatment Sequence 1 (Experimental): Subjects will receive two 75 mg micronized HPMC capsules, dosed fasted (Regimen C) in Period 1 and two 75 mg micronized HPMC capsules, dosed with a high-fat meal (Regimen D) in Period 2. Dosing will occur in the morning of Day 1 in each period, and dosing between periods will be separated by at least one week.
  Interventions: Drug: Regimen C; Drug: Regimen D
- Cohort 2 Treatment Sequence 2 (Experimental): Subjects will receive two 75 mg micronized HPMC capsules, dosed with a high-fat meal (Regimen D) in Period 1 and two 75 mg micronized HPMC capsules, dosed fasted (Regimen C) in Period 2. Dosing will occur in the morning of Day 1 in each period, and dosing between periods will be separated by at least one week.
  Interventions: Drug: Regimen C; Drug: Regimen D

INTERVENTIONS:
Drug: Regimen A — Two gelatin capsules containing 75 mg GSK2118436A (dosed as the mesylate salt, micronized particles, equivalent to 150 mg free base), dosed fasted
  Arms: Cohort 1 Treatment Sequence 1; Cohort 1 Treatment Sequence 2
Drug: Regimen B — Two gelatin capsules containing 75 mg GSK2118436A (dosed as the mesylate salt, larger, non-micronized particles, equivalent to 150 mg free base), dosed fasted
  Arms: Cohort 1 Treatment Sequence 1; Cohort 1 Treatment Sequence 2
Drug: Regimen C — Two Hydroxy Propyl Methyl Cellulose (HPMC) capsules containing 75 mg GSK2118436A (dosed as the mesylate salt, micronized particles, equivalent to 150 mg free base), dosed fasted
  Arms: Cohort 2 Treatment Sequence 1; Cohort 2 Treatment Sequence 2
Drug: Regimen D — Two HPMC capsules containing 75 mg GSK2118436A (dosed as the mesylate salt, micronized particles, equivalent to 150 mg free base), dosed with a high-fat meal
  Arms: Cohort 2 Treatment Sequence 1; Cohort 2 Treatment Sequence 2

SUMMARY:
The study is designed to evaluate the effects of a high fat meal on the pharmacokinetics of 150 mg of GSK2118436, as well as the effects of particle size on the relative bioavailability of GSK2118436.

DETAILED DESCRIPTION:
GSK2118436 is an orally administered, potent and selective small molecule BRAF inhibitor that is currently being developed for the treatment of BRAF mutation-positive tumors. This study is designed to evaluate the effects of particle size on the relative bioavailability of GSK2118436 (Cohort 1) and to evaluate the effects of a high-fat meal on the pharmacokinetics of GSK2118436 (Cohort 2). Subjects will randomly receive two of four possible regimens over two periods. Subjects enrolled in Cohort 1 will receive a single 150 mg dose of GSK2118436 as micronized particles fasted (gelatin capsule formulation) and a single 150 mg dose of GSK2118436 as non-micronized particles fasted (larger particle size). Subjects enrolled in Cohort 2 will receive a single 150 mg dose of GSK2118436 (HydroxyPropyl Methyl Cellulose (HPMC) capsule formulation) fasted and with a high-fat breakfast. GSK2118436 will be administered as the mesylate salt (equivalent to 150 mg free base). Safety and tolerability will also be evaluated. The study will be conducted at a sufficient number of centers to complete approximately 28 adult subjects (14 subjects per cohort) with BRAF mutation-positive tumors. Following completion of this study, subjects may continue dosing with GSK2118436 in the roll-over study, Protocol BRF114144.

ELIGIBILITY:
Inclusion Criteria:

* Male or female at least 18 years of age at the time of signing the informed consent form;
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form;
* Body weight >/= to 45 kg and a Body Mass Index (BMI) >/= to 19 kg/m2 and less than or equal to 35 kg/m2 (inclusive);
* Able to swallow and retain oral medication;
* BRAF mutation-positive tumor as determined via relevant genetic testing;
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1 at the time of transition to this study. NOTE: Subjects with an ECOG performance status of </= to 2 may be eligible with the approval of the GlaxoSmithKline (GSK) Medical Monitor.
* Women of child-bearing potential and men with reproductive potential must be willing to practice acceptable methods of birth control. Additionally, women of child-bearing potential must have a negative serum pregnancy test within 14 days prior to the first dose of study treatment;
* Must have adequate organ function as defined by the following values:
* Absolute neutrophil count (ANC) >/= to 1.2 x 10^9/L
* Hemoglobin >/= to 9 g/dL
* Platelets >/= to 100 x 10^9/L
* Serum bilirubin </= to 1.5 x upper limit of normal (ULN)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) </= to 2.5 x ULN; <5 x ULN if liver metastases are present (with approval of GSK medical monitor)
* Serum creatinine </= to ULN or calculated creatinine clearance >/= 60 mL/min
* Prothrombin time (PT)/International normalized ratio (INR) and partial thromboplastin time (PTT) < /= to 1.3 x ULN
* Left ventricular ejection fraction (LVEF) >/= to institutional lower limit of normal by Echocardiogram

Exclusion Criteria:

* Currently receiving cancer therapy (e.g., chemotherapy with delayed toxicity, extensive radiation therapy, immunotherapy, biologic therapy) within the last three weeks; chemotherapy regimens without delayed toxicity within the last two weeks; or use of an investigational anti-cancer drug within 28 days preceding the first dose of GSK2118436;
* Current use of a prohibited medication or requires any of these medications during the study;
* Consumption of red wine, Seville oranges, grapefruit or grapefruit juice from seven days prior to the first dose of study medication;
* Current use of therapeutic warfarin (note: low molecular weight heparin and prophylactic low-dose warfarin are permitted);
* History of sensitivity to heparin or heparin-induced thrombocytopenia;
* Any major surgery within the last four weeks;
* Unresolved toxicity greater than National Cancer Institute Common Terminology Criteria for Adverse Events, version 4.0 (NCI CTCAE v4.0) [NCI, 2009] Grade 2 from previous anti-cancer therapy except alopecia;
* Presence of active gastrointestinal disease or other condition (e.g., small bowel or large bowel resection) that will interfere significantly with the absorption of drugs. If clarification is needed as to whether a condition will significantly affect absorption of drugs, contact the GSK medical monitor for permission to enroll the subject;
* A history of known Human Immunodeficiency Virus (HIV), Hepatitis B Virus (HBV), or Hepatitis C Virus (HCV) infection (subjects with laboratory evidence of HBV clearance may be enrolled with permission of the GSK medical monitor);
* Presence of invasive malignancy other than one of the malignancies covered under Inclusion Criterion #5; patients with a history of malignancy that have been definitively treated can be enrolled with approval of the GSK medical monitor;
* Subjects with brain metastases are excluded if their brain metastases are either:

Symptomatic Treated (surgery, radiation therapy) but not clinically and radiographically stable one month after local therapy, or Asymptomatic and untreated but > 1 cm in the longest dimension Patients with small (≤ 1 cm in the longest dimension), asymptomatic brain metastases that do not need immediate local therapy can be enrolled with the approval of the GSK medical monitor. Subjects on a stable dose of corticosteroids for more than one month, or those who have been off corticosteroids for at least two weeks can be enrolled with approval of the GSK medical monitor. Subjects must also be off of enzyme-inducing anticonvulsants for more than four weeks;

* Presence of rheumatoid arthritis;
* History of alcohol or drug abuse within six months prior to screening;
* Corrected QT (QTc) interval >/= to 480 msecs;
* History of acute coronary syndromes (including unstable angina), coronary angioplasty, or stenting within the past 24 weeks;
* Class II, III, or IV heart failure as defined by the New York Heart Association (NYHA) functional classification system; abnormal cardiac valve morphology documented by echocardiogram (subjects with minimal abnormalities [ie, mild regurgitation/stenosis] can be entered on study with approval from the GSK medical monitor); or history of known cardiac arrhythmias (except sinus arrhythmias) within the past 24 weeks;
* Known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to the study drugs, or excipients (note: to date there are no known drugs chemically related to GSK2118436 which are approved by the Food and Drug Administration);
* Uncontrolled medical conditions (e.g., diabetes mellitus, hypertension), psychological, familial, sociological, or geographical conditions that do not permit compliance with the protocol; or unwillingness or inability to follow the procedures required in the protocol;
* Subjects with known glucose 6 phosphate dehydrogenase (G6PD) deficiency;
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, five half-lives or twice the duration of the biological effect of the investigational product (whichever is longer);
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period;
* Pregnant females as determined by positive human chorionic gonadotrophin (hCG) test at screening or prior to dosing;
* Lactating females who are actively breast feeding;
* Subject is mentally or legally incapacitated;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2010-10-21 (Actual); Primary Completion 2011-05-13 (Actual); Study Completion 2011-05-13 (Actual)

PRIMARY OUTCOMES:
Area under the plasma-concentration time curve (AUC) of GSK2118436 | 0, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 24, 48, 72 and 96 hours post-dose
Maximum plasma concentration (Cmax) of GSK2118436 | 0, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 24, 48, 72 and 96 hours post-dose
Time to Cmax (Tmax) of GSK2118436 | 0, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 24, 48, 72 and 96 hours post-dose

SECONDARY OUTCOMES:
Terminal half-life (t1/2) of GSK2118436 | 0, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 24, 48, 72 and 96 hours post-dose
AUC, Cmax, Tmax and t1/2 of GSK2118436 metabolites (GSK2285403, GSK2167542 and GSK2298683) and ratio of metabolite to parent drug GSK2118436 | 0, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 24, 48, 72 and 96 hours post-dose
Number of subjects with adverse events as a measure of safety and tolerability | From date of first dose until transition to rollover protocol BRF114144 (approximately 12 days) or study follow up visit if subject does not transition to BRF114144 (approx 22 days)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (4):
- United States (4):
  - GSK Investigational Site, Scottsdale, Arizona
  - GSK Investigational Site, Detroit, Michigan
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, Salt Lake City, Utah

REFERENCES:
- [Derived] Ouellet D, Grossmann KF, Limentani G, Nebot N, Lan K, Knowles L, Gordon MS, Sharma S, Infante JR, Lorusso PM, Pande G, Krachey EC, Blackman SC, Carson SW. Effects of particle size, food, and capsule shell composition on the oral bioavailability of dabrafenib, a BRAF inhibitor, in patients with BRAF mutation-positive tumors. J Pharm Sci. 2013 Sep;102(9):3100-9. doi: 10.1002/jps.23519. Epub 2013 Apr 22. PMID 23608920
- See also: Results for study 113468 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/113468?search=study&study_ids=113468#rs